CLINICAL TRIAL: NCT07276724
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of GB-0895 Adjunctive Therapy in Adults and Adolescents With Severe Uncontrolled Asthma
Brief Title: A Study to Investigate GB-0895 Adjunctive Therapy in Adults and Adolescents With Severe Uncontrolled Asthma (SOLAIRIA-1)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Generate Biomedicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GB-0895-301 (SOLAIRIA-1)
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Severe Asthma
Keywords: Asthma; Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GB-0895 (Experimental): GB-0895 Subcutaneous (SC) injection
  Interventions: Drug: GB-0895
- Placebo (Placebo Comparator): Placebo Subcutaneous (SC) injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GB-0895 — Study Drug
  Arms: GB-0895
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the potential for GB-0895 treatment to improve the health of adolescents and adults with severe asthma that is uncontrolled by inhaled corticosteroids (ICS) and conventional asthma controllers.

The study details include:

Study treatment: randomized to receive either GB-0895 or placebo administered every 6 months over 52 weeks.

Visit frequency: every 1-2 months after the first month.

DETAILED DESCRIPTION:
This is a global, multicenter, randomized, double-blind, placebo-controlled Phase 3 study to evaluate the efficacy and safety of GB-0895 adjunctive therapy in adults and adolescents with severe uncontrolled asthma with an optional open-label extension (OLE). The trial is designed to administer GB-0895 an investigational drug or placebo, subcutaneously every 6 months.

The study is divided into several phases as described below:

* Screening/Baseline (Weeks -6 to -4)
* Run-in (Weeks -4 to 0, ±1)
* Treatment (Weeks 0 to 52)
* Follow-up (Weeks 52 to 90) or optional open-label extension (OLE) (Weeks 52 to 142, OLE includes GB-0895 treatment on Week 52 and Week 78)

Approximately 786 eligible study participants will be screened and randomized globally to receive either GB-0895 or placebo at week 0 and week 26. The safety of the participants enrolled in this trial will be carefully monitored.

ELIGIBILITY:
1. Adults and adolescents ≥ 12 and ≤ 80 years of age.
2. Documented physician diagnosis of asthma for ≥ 2 years.
3. Subjects must be on medium to high dose ICS for ≥ 12 months before Screening Visit 1 plus at least 1 additional asthma controller (e.g., LABA, LAMA) ≥ 3 months before Screening Visit 1 with no change in ICS or controller(s) for at least three months.
4. Subjects must have a well-documented history of at least two asthma exacerbations requiring systemic corticosteroid treatment despite the use of medium-to-high dose ICS in the past 12 months before Screening Visit 1.
5. Adults ≥ 18 years of age at Screening Visit 1, a pre-BD FEV1 <80% predicted at Screening Visit 1.
6. Adolescents 12 to < 18 years of age at Screening Visit 1: A pre-BD FEV1 < 90% predicted OR, FEV1:Forced Vital Capacity (FVC) ratio < 0.80.
7. Positive BD responsiveness test: Increase of at least 12% and 200 mL in FEV1 between 15 and 60 minutes after the administration of a short-acting β2-agonist (SABA) at least once during the screening period.
8. ACQ-6 score ≥ 1.5 at the Screening Visit.
9. Weight ≥40 kg at the Screening Visit 1

Exclusion Criteria:

1. Subjects who experience a clinically significant asthma exacerbation within 12 weeks before the Screening Visit or during the run-in period and require a change in asthma maintenance therapy.
2. Other concurrent respiratory disease other than asthma, including (but not limited to) current infection, bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis, tuberculosis, diagnosis of chronic pulmonary disease (including but not limited to emphysema and/or chronic bronchitis), or a history of lung cancer.
3. Eosinophilic disease (e.g., eosinophilic granulomatosis with polyangiitis, eosinophilic esophagitis).
4. Any cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could affect subject safety, influence study findings or interpretation, or impede completion of the study.
5. Clinically significant infection that is unresolved and requires systemic antibiotic, antifungal, antiparasitic, or antiviral medications preceding enrollment.
6. A current malignancy or previous history of cancer within 5 years before screening.
7. Clinically significant infection that is not resolved before study enrollment.
8. Subjects with a known, pre-existing helminth parasitic infestation within 6 months before Screening Visit 1.
9. Current smokers or subjects with a smoking history ≥10 pack-years, and subjects using vaping products, including electronic cigarettes.
10. Former smokers with a smoking history of <10 pack-years and users of vaping/e-cigarette products must have stopped for at least 6 months before Screening Visit 1 to be eligible.
11. Hepatitis B, C, or HIV.
12. Major surgery within 8 weeks before Screening Visit 1 or planned surgical procedures requiring general anesthesia or inpatient status for >1 day during the study.
13. Use of any anti-IL-5 therapy (e.g., mepolizumab, reslizumab, benralizumab, depemokimab) within 12 months before Screening Visit 1 or other monoclonal antibodies used for asthma within 4 months or 5 half-lives.
14. Prior use (at any time) of any anti-TSLP or anti-TSLP receptor biologics, approved (e.g., tezepelumab) or investigational.
15. Treatment with systemic immunosuppressive/immunomodulating drugs (e.g., methotrexate, cyclosporine) within 12 weeks prior to randomization.
16. Receipt of an investigational biologic within 4 months or 5 half-lives, OR receipt of an investigational non-biologic within 30 days or 5 half-lives before Screening Visit 1.
17. Known history of sensitivity to any component of the study treatment formulation.
18. History of life-threatening anaphylaxis following any biologic therapy.
19. Concurrent enrollment in another clinical study involving investigational product (IP).
20. Subject has been randomized in the current study or previous GB-0895 studies.
21. Any clinically meaningful abnormal finding in physical examination, vital signs, ECG, hematology, serum chemistry, or urinalysis that, in the opinion of the Investigator, may put the subject at risk, influence study results, or impede study completion.
22. Cirrhosis (with or without hepatic dysfunction) or other active or clinically significant liver disease.
23. Receipt of immunoglobulin or blood products within 30 days before Screening Visit 1.
24. Receipt of live attenuated vaccines within 30 days before randomization and during the study, including the follow-up period.
25. Receipt of the T2 cytokine inhibitor suplatast tosilate within 15 days before Screening Visit 1.
26. Subjects treated with bronchial thermoplasty in the last 12 months before Screening Visit 1.
27. Unwillingness or inability to follow study procedures, including poor adherence to asthma controller medications, in the opinion of the Investigator.
28. Women who are pregnant, lactating, or planning to become pregnant during the study.
29. History (or suspected history) of alcohol misuse or substance abuse within 2 years before Screening Visit 1.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 786 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the annualized asthma exacerbation rate (AAER) in adult and adolescent subjects with severe uncontrolled asthma. | From Day 1 (randomization) to Week 52
  The annual exacerbation rate is based on clinically significant (CS) exacerbations reported by the investigator in the electronic case (eCRF) over 52 weeks for subjects on GB-0895 as compared to placebo.

SECONDARY OUTCOMES:
To evaluate the annualized asthma exacerbation rate (AAER) in adult and adolescent subjects with severe uncontrolled asthma and baseline eosinophils (EOS) < 300 cells/µL. | From Day 1 (randomization) to Week 52
  The annual exacerbation rate is based on CS exacerbations reported by the investigator in the eCRF over 52 weeks for subjects with baseline EOS < 300 cells/ µL on GB-0895 as compared to placebo.
Change from baseline in pre-bronchodilator (BD) forced expiratory volume in 1 second (FEV1) | From Day 1 (randomization) to Study Week 52
  The change from baseline in pre-BD FEV1 for subjects on GB-0895 as compared to placebo at week 52. FEV1 is defined as the volume of air exhaled from the lungs in the first second of a forced expiration.
Change from baseline in Asthma Quality of Life Questionnaire AQLQ(S)12+ score | From Day 1 (randomization) to Week 52
  The change from baseline on AQLQ(S)12+ score for subjects on GB-0895 as compared to placebo at week 52. The AQLQ(S)12+ is a 32-question assessment with questions related to symptoms, activity limitations, emotional function, and environmental stimuli. Questions are scored on a 7-point scale, which ranges from 7 (no impairment) to 1 (severe impairment). The overall score is calculated as the mean to all questions.
Change from baseline in Asthma Control Questionnaire (ACQ-6) score | From Day 1 (randomization) to Week 52
  The change from baseline on ACQ-6 score for subjects on GB-0895 as compared to placebo at week 52. The ACQ-6 is a 6-question questionnaire that assesses asthma symptoms (e.g., activity limitation, shortness of breath, wheezing etc.). Questions are scored on a 6-point scale, where 0 corresponds to totally controlled asthma and 6 corresponds to severely uncontrolled asthma.
Time to first asthma exacerbation from randomization | From Day 1 (randomization) to Week 52
  After subjects complete the screening period and are randomized to either GB-0895 or placebo, the time it takes until the first clinically significant asthma exacerbation occurs. Clinically significant asthma exacerbations are defined as requiring systemic corticosteroids (oral, IV, or intramuscular) and/or hospitalization or emergency department visits requiring systemic corticosteroids.
Change from baseline in weekly mean daily Asthma Daytime Symptom Diary (ADSD) | From Day 1 (randomization) to Week 52
  The change from baseline on weekly mean daily ADSD score for subjects on GB-0895 as compared to placebo at week 52. The ADSD is an 8-question diary that assesses asthma symptoms that the subjects will fill out at night before bed.
  The ADSD daily score is calculated by averaging the 8 daily score and a mean of 7-day ADSD score is calculated by averaging of the 7 daily score. The daily score is not calculated if any item response is missing.
Change from baseline in weekly mean daily Asthma Nighttime Symptom (ANSD) | From Day 1 (randomization) to Week 52
  The change from baseline on daily ANSD score for subjects on GB-0895 as compared to placebo at week 52.
  ANSD is an eight-question diary that assesses asthma symptoms that the subjects will fill out in the morning upon waking. The ANSD score is calculated by averaging the 8 daily score and a mean of 7-day ANSD score is calculated by averaging of the seven daily score.
Change from baseline in St. George's Respiratory Questionnaire (SGRQ) total score | From Day 1 (randomization) to Week 52
  The change from baseline on SGRQ score for subjects on GB-0895 as compared to placebo at week 52. The SGRQ is a 50-item questionnaire designed to measure health status. Questions are scored on a range of 0 to 100, with a lower score indicating a better quality of life
Change from baseline in 22-Item Sino-Nasal Outcomes Test (SNOT-22) score | From Day 1 (randomization) to Week 52
  The change from baseline on SNOT-22 score for subjects on GB-0895 as compared to placebo at week 52.The SNOT-22 is a 22-question questionnaire that assesses the impact on health-related quality of life and questions are scored from 0 to 110, with 0 indicating no disease and 110 as the worst disease.
Change from baseline in the 5-Level EuroQol 5 dimensions questionnaire (EQ-5D-5L) score | From Day 1 (randomization) to Week 52
  The change from baseline on EQ-5D-5L score for subjects on GB-0895 as compared to placebo at week 52. The EQ-5D-5L questionnaire includes a visual analogue scale (VAS) that allows subjects to rate current health status on a 0-100 scale, with 0 being the worst imaginable health state.
PGI-S response at Week 52 | From Day 1 (randomization) to Week 52
  The Patient Global Impression of Asthma Severity (PGI-S) at Week 52 defined as an improvement by 1 or more points on the 0-5 scale. The PGI-S questionnaire asks the subjects to rate the overall severity of their asthma symptoms of the past 7 days with response options of: 1= no asthma symptoms, 2= mild, 3= moderate, 4= severe, and 5= worst possible asthma symptoms.
ACQ-6 response at Week 52 | From Day 1 (randomization) to Week 52
  The Asthma Control Questionnaire-6 (ACQ-6) at Week 52 defined as an improvement in score of 0.5 or more.
  The ACQ-6 questionnaire is a 6-question subject-reported questionnaire that assesses the most common asthma symptoms and responses are calculated from the mean of the scores out of a value of 6, where 0 corresponds to totally controlled asthma and 6 corresponds to severely uncontrolled asthma.
AQLQ(S)12+ response at Week 52 | From Day 1 (randomization) to Week 52
  The Asthma Quality of Life Questionnaire for 12-Year-Old and Older at week 52 defined as an improvement in score of 0.5 or more. The AQLQ(S)12+ is a 32-question subject-reported assessment. The questions are scored on a 7-point scale, which ranges from 7 (no impairment) to 1 (severe impairment). The overall score is calculated as the mean of all questions.
SGRQ response at Week 52 | From Day 1 (randomization) to Week 52
  The St. George's Respiratory Questionnaire at week 52 defined as achieving ≥ 4-point reduction from baseline. The SGRQ is a 50-item questionnaire designed to measure health status and questions are scored on a range of 0 to 100, with a lower score indicating a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Snodgres, Study Director — Generate Biomedicines
Locations (1):
- Research Site 01, Miami Lakes, Florida, United States